CLINICAL TRIAL: NCT03294889
Title: ONE-SHOT - Single Shot Radiotherapy for Localized Prostate Cancer. A Multicenter, Single Arm, Phase I/II Trial
Brief Title: ONE-SHOT Trial - Ultra-hypofractionated Single-dose SBRT for Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: Humanitas Hospital, Italy (Other); University of Zurich (Other); Kantonsspital Graubünden (Other)
Responsible Party: Principal Investigator, Thomas Zilli, Médecin Adjoint Agrégé, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-01236
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Stereotactic body radiation therapy; Calypso® beacon system
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Stereotactic body radition (SBRT) — Ultra-hypofractionated single-fraction SBRT with urethra-sparing with image-guidance and intra-fractional control motion with the Calypso® system.
  * 19 Gy in a single fraction to the whole prostate gland ± proximal seminal vesicles
  * 17 Gy in a single fraction to the urethra planning-risk volume (PRV)

SUMMARY:
The main objective of the phase I/II trial is to determine the safety and efficacy of a single fraction SBRT at a dose of 19 Gy in patients with localized prostate cancer.

DETAILED DESCRIPTION:
Total dose and dose per fraction play an important role in the curative treatment of prostate cancer with radiotherapy (RT). Modern image guided external RT allows safe dose escalation of prostate cancer. There are strong radiobiological and clinical considerations that suggest that treatment with a small number of large fractions (hypofractionation) may increase the therapeutic ratio of RT for prostate cancer by increasing the tumor cell killing effect with relatively less toxic effect on the surrounding late responding normal tissues compared to conventional fractionation.

The question of how far can the number of fractions with SBRT be reduced is an exciting research matter with an undoubtful goal, face the challenge of assessing the potential for cure of prostate cancer patients with a single and unique fraction of high dose irradiation similar to what is already undertaken with radiosurgery against brain, lung, and liver targets.

We hypothesize that an ultra-hypofractionated single-dose SBRT employing state of the art of image-guided RT techniques may be feasible, with a safe toxicity profile and an optimal long-term tumor control. Hence, a prospective phase I/II clinical trial will be initiated in prostate cancer patients with a localized disease to validate this treatment schedule as an alternative to normofractionated/moderate hypofractionated RT schedules to be tested in a second time in a phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent according to ICH/GCP regulations before registration and prior to any trial specific procedures
* Histologically confirmed adenocarcinoma of the prostate without small cell features
* Tumor clinical stage cT1c-2c, pN0 or cN0, M0, according to UICC TNM 2009
* MRI staging must confirm American Joint Committee on Cancer (AJCC) stage T1, T2a, T2b or T2c
* Gleason score at biopsy 3+3 or 3+4 (WHO 2016 Grade Groups 1, 2)
* PSA ≤15 ng/ml
* WHO performance status 0-1
* International Prostate Symptom Score ≤ 10 (alpha blockers allowed)
* MRI-based volume estimation of prostate gland ≤ 70 cc
* Patient agrees not to father a child during trial treatment and during 6 months thereafter

Exclusion Criteria:

* Tumor clinical stage cT3a-3b or T4
* Evidence of T3a, T3b or T4 disease as assessed by MRI
* Positive lymph-nodes or metastatic disease from prostate cancer on imaging studies.
* Significant tumor on the transitional zone as assessed by MRI
* Gleason at biopsy ≥ 4+3
* Androgen deprivation therapy or products known to affect PSA levels
* Impossibility to implant Calypso beacons
* History of hematologic or primary solid tumor malignancy, unless in remission for at least 3 years from registration with the exception of curatively treated localized non-melanoma skin cancer
* Prior pelvic radiotherapy
* Previous surgery for prostate cancer
* Previous transurethral resection of the prostate (TURP) (< 12 weeks before registration)
* Hip prosthesis
* Severe or active co-morbidity likely to impact on the advisability of SBRT
* Any other serious underlying medical, psychiatric, psychological, familial or geographical condition, which in the judgment of the investigator may interfere with the planned staging, treatment and follow-up, affect patient compliance or place the patient at high risk from treatment-related complications

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Histologically confirmed adenocarcinoma of the prostate
Enrollment: 45 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | 3 months
  Toxicity will be evaluated using Grade ≥ 3 genitourinary and/or gastrointestinal acute adverse event (AE) during the first 3 month according to CTCAE classification v.4.03 (Phase I).
Progression free survival (PFS) | 3 years
  The primary endpoint is 3-years biochemical relapse free survival (bRFS). bRFS and its 97.5% one-sided confidence interval (CI) will be determined using the Kaplan Meier method. If the expected value of 96% isn't included in this interval, the efficacy of the experimental treatment will be questioned. (Phase II).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Zilli, MD, Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zilli T, Scorsetti M, Zwahlen D, Franzese C, Forster R, Giaj-Levra N, Koutsouvelis N, Bertaut A, Zimmermann M, D'Agostino GR, Alongi F, Guckenberger M, Miralbell R. ONE SHOT - single shot radiotherapy for localized prostate cancer: study protocol of a single arm, multicenter phase I/II trial. Radiat Oncol. 2018 Sep 4;13(1):166. doi: 10.1186/s13014-018-1112-0. PMID 30180867